CLINICAL TRIAL: NCT02339467
Title: Getting Older Adults OUT-of-doors (GO-OUT): A Randomized Controlled Trial of a Community-based Outdoor Walking Program
Brief Title: Getting Older Adults OUT-of -Doors
Acronym: GO-OUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Toronto (Other); McGill University (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2014:391
Record Dates: First submitted 2015-01-07; First posted 2015-01-15 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2016-05

CONDITIONS: Older Adults With Decreased Outdoor Walking Ability
Keywords: decreased outdoor walking ability; Older adult

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GO-OUT program (Experimental): An outdoor walking workshop with stations to learn various outdoor walking skills and information, followed by a supervised, group based outdoor walking program, twice a week for 60 minutes, for 3 months.
  Interventions: Other: GO-OUT program
- Task-oriented outdoor walking workshop (Active Comparator): An outdoor walking workshop with stations to learn various outdoor walking skills and information.
  Interventions: Other: Task-oriented outdoor walking workshop

INTERVENTIONS:
Other: GO-OUT program — Participants attend the walking workshop followed by a 3-month outdoor walking group intervention, twice weekly for 60-minutes. Each session includes a 10-minute warm-up and cool down, and a planned walk in an outdoor community environment. Continuous walking exercise will gradually increase from 10 to 60 minutes, as well increase difficulty. Balance exercises will be included in the warmup and walk. There will be a variety of surfaces and environmental factors to challenge the participants, e.g., carrying objects, diverting the walker's attention, crossing at a light, walking up and down curbs, slopes, and level or uneven surfaces. Supervision will be on a 1:3 facilitator-to-participant ratio to allow for assistance and individualization of the intervention where necessary.
  Arms: GO-OUT program
Other: Task-oriented outdoor walking workshop — The 1-day workshop will be 5 hours with breaks. Participants will complete a series of stations learning information, strategies and skills related to safely walking outdoors. Stations include: pedometer use; walking pole use; footwear; footcare; fall prevention; balance exercises; proper use of walking aids; correct posture; self-management of exercise intensity; goal setting; and walking safely outdoors. Participants will receive a workbook with Canadian Physical Activity Guidelines, benefits of outdoor walking, information for each workshop station and a pedometer. Participants will use the workbook as an information resource and to record their community ambulation goals, planning routes, and walking time. All participants will be encouraged to walk outside with a partner, for safety.
  Arms: Task-oriented outdoor walking workshop

SUMMARY:
Community walking is an issue that older adults with chronic conditions have described as important to participation in the community. Walking outside the home is a universally accessible form of physical activity that has multiple health benefits. Walking for 150 minutes per week can help reduce the risk of cardiovascular disease, hypertension, stroke, diabetes, osteoporosis, and depression, as well as falls. Practice walking across roads, slopes and curbs, while talking, and dealing with crowds and traffic, is safe and feasible and can improve confidence, balance and walking ability. Being physically active outdoors in nature appears to improve mental health more than being active indoors. Despite these health benefits, the majority of older Canadians do not walk outside on a regular basis. Barriers to walking outside include fear, physical disability due to chronic disease, the appropriateness of footwear and walking aids, and the physical environment, such as uneven pavement, weather and temperature. To date, the best strategy for getting people to walk outdoors regularly is unknown. The investigators propose to evaluate the effectiveness of a dynamic 1-day workshop, at which older adults who infrequently walk outdoors learn strategies to facilitate outdoor walking, such as appropriate use of footwear, ambulatory aids and equipment, goal setting, and practice skills related to increasing outdoor walking. The workshop will be compared to the workshop plus involvement in a walking group for 3 months. Outcomes include outdoor walking activity, total physical activity, walking ability, participation, and health-related quality of life. Each participant will have three evaluations: before the intervention and 3 and 6 months later. The investigators will interview select participants at 6 months to ask them about their opinions of what worked and didn't work. Increasing outdoor walking is expected to improve health and well-being, and help people live independently in the community for longer.

DETAILED DESCRIPTION:
Background: Inability to walk outdoors restricts full participation in physical activity and community living for older adults that can reduce health-related quality of life (HRQL). Older adults report limited outdoor walking with only 8% achieving the Canadian recommendation for older adults of 150 minutes of moderate-to-vigorous (MV) intensity physical activity per week. Known barriers to walking outside include fear, physical disability due to chronic disease, the appropriateness of footwear and walking aids, the physical environment, weather and temperature. Group practice walking outdoors in locations with variable environmental challenges has the potential to improve physical ability, confidence, outdoor and overall physical activity and social participation. The extent to which it is safe and feasible to implement this intervention in people with varying degrees of physical ability, preferences for where to walk, neighbourhood walkability, and to measure outdoor walking activity, is unclear.

Objectives: The study purpose is to evaluate the feasibility of a randomized controlled trial (RCT) protocol designed to evaluate the effectiveness of an education and skills workshop plus a 3-month outdoor walking group (GO-OUT program) compared to the workshop alone in improving outdoor walking activity. Specific objectives are to characterize participants; determine the feasibility of recruitment; estimate withdrawal rates and the safety and feasibility of the study protocol; obtain preliminary effect sizes; identify the optimal measure of outdoor walking activity based on validity, reliability, effect size and data completeness; and identify participants' and intervention facilitators' perceptions of the challenges and benefits of the intervention and evaluation tools.

Methods: Design and Participants-A feasibility RCT with an embedded qualitative component is proposed with 18 participants. Ambulatory older adults living in the community who report walking outdoors ≤20 minutes/week will be stratified by level of walking impairment (gait speed<0.8 m/s vs ≥0.8 m/s) and randomly assigned to receive the GO-OUT program or the workshop alone. Group allocation will be concealed. A blinded evaluator will evaluate participants at baseline, 3 and 6 months. At 6 months, focus groups of participants from the GO-OUT and workshop groups and intervention facilitators, will participate in a semi-structured interview to explore perceived benefits and challenges of adherence, intervention strategy and outcome measures. Interventions-The workshop will include activity stations at which people will learn about appropriate footwear, walking aids and equipment (pedometers, Nordic poles), goal setting, physical activity recommendations/benefits and practice walking-related tasks. The GO-OUT program will include the workshop plus the outdoor walking group. The walking group will be supervised and consist of 9 participants; they will meet twice a week for 1 hour to walk in increasingly challenging environments to achieve individualized goals. Outcome Measures-Outdoor walking (primary outcome) will be measured by 2 methods: outdoor walking items of the Community Health Activities Model Program for Seniors (CHAMPS) (self-report) and accelerometer/Global Positioning System (GPS). Overall physical activity (secondary outcome) will be measured with the CHAMPS (self-report) as well as accelerometry. Measures of aerobic capacity, walking competency, mood, participation, and HRQL will also be administered. Neighbourhood walkability will be assessed with the Neighbourhood Environment Walkability Scale (self-report). Analysis-This is a feasibility study; therefore, no hypotheses will be tested. The analysis will include describing participant characteristics, estimating recruitment, withdrawal and adverse event rates, estimating preliminary effect sizes for outcome measures, estimating test-retest reliability of outdoor walk time derived from the CHAMPS and construct validity and data completeness of outdoor walk time derived from the CHAMPS and accelerometry/GPS. A qualitative descriptive approach will be used to analyse the interview data. Conclusion-Increasing outdoor walking is expected to help people improve physical activity, the ability to live independently in the community, and health and well-being. This study will evaluate the feasibility of a trial protocol aimed at improving outdoor walking. Findings will be used to justify and inform planning of a future definitive multi-site trial.

ELIGIBILITY:
Inclusion Criteria:

* self-reported ability to walk continuously on a flat surface a distance of ≥1 block (~50 metres or 164 feet) independently with or without a walking aid and without supervision
* outdoor walking limitation defined as self-reportedly accumulating ≤20 minutes of outdoor walking in a typical week
* mental competency indicated by a score of ≥18 on the telephone version of the Mini-mental State Exam

Exclusion Criteria:

* active walkers defined as accumulating ≥100 minutes of total (indoor and outdoor) walking per week
* have had ≥2 falls in the prior 12 months or present with an acute fall (based on American Geriatric Society fall guidelines)
* cardiac, respiratory, peripheral vascular or other health conditions that would prevent safe and full participation in the interventions
* currently receiving rehabilitation treatment such as physical or occupational therapy for goals related to walking
* postural hypotension determined by measuring lying and standing blood pressure
* severe limitations to visual acuity by a falls prevention screen
* resting heart rate under 45 or over 100.

The PAR-Q+ (an evaluation of exercise readiness) will be completed by each participant. With participants' permission, their family physician will be asked to review the PAR-Q+ and confirm readiness to participate in exercise.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Outdoor walking activity - CHAMPS questionnaire | baseline, 3,6 months
  Self-report measure designed to evaluate interventions to increase physical activity among older persons. Will determine number of minutes at moderate to vigorous intensity of walking outdoors per week by focusing on 4 walking items.
Change in Outdoor walking activity -GPS data | baseline, 3,6 months
  Participants will wear the GlobalSat DG-200 Data Logger (www.gpscentral.ca/products/usglobalsat/dg200.html) clipped onto their waist band from the time they first get out of bed in the morning until they return to bed in the evening, removing it for showering, bathing, and swimming, for 14 days. Will determine The number of minutes spent walking per week outdoors.
Change in Outdoor walking activity -Accelerometry | baseline, 3,6 months
  The ActiGraph GT3X+ monitor (www.actigraphcorp.com/products/wgt3x-monitor/, ActiGraph, Pensacola, FL) will be worn by each participant, clipped onto their waist band over the right hip on the anterior axillary line along with the GPS. Time spent in sedentary, light, moderate and high intensity PA categories/day will be calculated.

SECONDARY OUTCOMES:
Change in Aerobic capacity (Six minute walk test) | baseline, 3,6 months
  Six minute walk test - distance walked in 6 minutes.
Change in Walking competency (Berg Balance scale) | baseline, 3,6 months
  Balance, lower limb strength, ambulation self-efficacy, and walking speed will be evaluated using the Berg Balance scale, the sit to stand test, the Ambulation Self-efficacy Scale, and the 10-metre walk test (gait speed), respectively.
Change in Mood (Geriatric depression scale) | baseline, 3,6 months
  Geriatric depression scale. If a participant scores >9, they will not be excluded, but the family physician will be notified.
Change in Health Related Quality of life (The Rand-36) | baseline, 3,6 months
  The Rand-36, self reported mental health and physical function.
Change in Participation (CHAMPS) | baseline, 3,6 months
  Time in minutes per week spent performing all 40 social, leisure and physical activities described in the CHAMPS will be used in the analysis.

OTHER OUTCOMES:
Neighbourhood walkability (Neighbourhood Environment Walkability Scale (NEWS) | baseline
  67-item self-report Neighbourhood Environment Walkability Scale (NEWS). Socio-economic characteristics of neighbourhoods in which participants reside will also be collected, using neighbourhood census data. NEWS is the most commonly internationally used self-report measure.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Barclay, PhD, Principal Investigator — University of Manitoba; Nancy Salbach, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Manitoba College of Rehabilitation Sciences, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Barclay R, Webber S, Ripat J, Grant T, Jones CA, Lix LM, Mayo N, van Ineveld C, Salbach NM. Safety and feasibility of an interactive workshop and facilitated outdoor walking group compared to a workshop alone in increasing outdoor walking activity among older adults: a pilot randomized controlled trial. Pilot Feasibility Stud. 2018 Nov 29;4:179. doi: 10.1186/s40814-018-0367-4. eCollection 2018. PMID 30519481